CLINICAL TRIAL: NCT03898856
Title: Yield of Diagnostic Tests and Management of Crofelemer for Chronic Idiopathic Diarrhea In Non-HIV Patients: A Pilot Study
Brief Title: Yield of Diagnostic Tests and Effects of Crofelemer for Chronic Idiopathic Diarrhea In Non-HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Brooks Cash, Visiting professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0990
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Diarrhea of Unknown Origin
Keywords: diarrhea; diagnosis; crofelemer; treatment
MeSH Terms: conditions — Diarrhea; Disease | interventions — crofelemer; Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crofelemer and Diagnostic tests for cause of chronic diarrhea (Experimental): 125 mg tablets taken by mouth twice daily for 28 days
  Interventions: Drug: Crofelemer; Diagnostic Test: Diagnostic tests for cause of chronic diarrhea

INTERVENTIONS:
Drug: Crofelemer — 125 mg tablets taken by mouth twice daily for 28 days
Diagnostic Test: Diagnostic tests for cause of chronic diarrhea — Diagnostic tests include: Esophagogastroduodenoscopy, Colonoscopy, biopsies of the upper gastrointestinal tract (duodenum) and lower gastrointestinal tract (colon), genetic testing for Congenital sucrase-isomaltase deficiency (CSID),Prometheus IBcause Chronic Diarrhea panel, Thyroid Panel, Stool osmolality, Stool Ova and Parasites, Stool Culture, Stool Qualitative Stool Fat, Stool Reducing Substances, Laxative Screening, Lactulose Hydrogen Breath Test, Gastrin Level, Calcitonin Level, Vasoactive Intestinal Polypeptide(VIP) level.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the drug Crofelemer in the treatment of non-HIV patients with chronic idiopathic diarrhea; to determine the prevalence of identifiable causes of chronic diarrhea in a non-HIV patients; to assess the diagnostic yield, in terms of identification of treatable etiologies, of commercially available diagnostic evaluations in adult, non-HIV patients with chronic idiopathic diarrhea, that is, evaluate which tests, among the standard diagnostic tests commonly conducted as part of the evaluation of chronic idiopathic diarrhea, are most likely to identify a treatable cause of the diarrhea; and to analyze the relationship between chronic idiopathic diarrhea and health-related quality of life and assess the impact of crofelemer treatment on health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic diarrhea (defined as 3 non-bloody loose stools per day or more than 20 non-bloody loose stools per week for more ≥ 4 weeks) and Bristol Stool Form Scale for stool consistency of 6/7 with >50% stool without an obvious cause after evaluation for organic etiologies.
* Patients from any ethnicity

Exclusion Criteria:

* Hematochezia (potentially related to an organic cause).
* Subjects less than 18 years of age more than 75 years of age (safety and effectiveness of crofelemer has not been established in these age groups).
* Pregnant females (crofelemer is a Category C drug due to lack of well-controlled studies to study its effects in this population).
* Lactating females (it is unknown if crofelemer is excreted in the human milk and thus may have unknown adverse effects on the nursing infants).
* HIV positive individuals.
* Persons within ability to provide consent and understand the study
* Persons with history of alcohol abuse or binge drinking.
* Persons with history of surgical bowel resection or bariatric surgery in the past 12 months.
* Persons who have undergone cholecystectomy (open or laparoscopic) in the past 3 months.
* Persons receiving antibiotics currently or have received antimicrobials in the past 4 weeks.
* Persons with end-organ failures including end-stage renal disease, end-stage liver disease, or severe heart failure.
* Persons with metastatic hematologic and oncologic malignancies.
* Persons receiving chemo-radiation or immune-modulators for oncologic or rheumatologic conditions.
* Persons with any other known organic gastrointestinal or non-gastrointestinal disease process in which diarrhea is a recognized clinical feature.
* Gluten free diet for previous 3 months and refusal to ingest gluten.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Cash, MD, Principal Investigator — The University of Texas Health Sciences Center at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 93 participants enrolled, 23 met the inclusion criteria and continued in the study to receive the intervention.
Period: Overall Study
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Started | 93
Received Intervention | 23
Completed | 23
Not Completed | 70

BASELINE CHARACTERISTICS:
Population: includes all participants who received the intervention
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 50 Percent Decrease in Mean Stool Count
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Participants | 17

2. Secondary Outcome: Number of Participants With an Improvement in Stool Consistency by More Than 2 Levels as Measured by the Bristol Stool Form Scale
Description: The Bristol stool form scale is a validated 1-7 scale that correlates to stool form. Type 1 is pebble like stool, type 2 lumpy and hard, type 3 like a sausage with cracks on the surface type 4 like a sausage but smooth and soft, type 5 soft blobs with clear cut edges, type 6 fluffy pieces with ragged edges, mushy stool, type 7watery, no solid pieces Types 5-7 are consistent with diarrhea and for this study a movement to lower types is considered an improvement
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Participants | 18

3. Secondary Outcome: Physical, Psychological, and Social Functioning as Measured by the Health-related Quality of Life (HRQOL) Questionnaire
Description: Health-related quality of life questionnaire assesses psychological, and social functioning. The total score ranges from 0 to 100 with higher scores indicate better quality of life.
Time Frame: Baseline,week 4 of treatment
Population: Data were only collected from participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 16
score on a scale
  Baseline | 63.8 (9.32)
  Week 4 | 61.8 (8.75)

4. Secondary Outcome: Number of Participants With Any Abnormal Diagnostic Test Results Leading to the Identification of the Cause of Chronic Diarrhea
Time Frame: Baseline
Population: Data were not collected for 5 participants because required laboratory assessments were not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 88
Participants | 12

5. Primary Outcome: Number of Participants With a 50 Percent Decrease in Mean Stool Count
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Participants | 16

6. Primary Outcome: Number of Participants With a 50 Percent Decrease in Mean Stool Count
Time Frame: Week 3
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Participants | 18

7. Primary Outcome: Number of Participants With a 50 Percent Decrease in Mean Stool Count
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
Number analyzed (Participants) | 23
Participants | 17

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Crofelemer and Diagnostic Tests for Cause of Chronic Diarrhea
All-Cause Mortality (participants affected / at risk) | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03898856/Prot_SAP_000.pdf